CLINICAL TRIAL: NCT03522519
Title: Profiling and Predicting the Natural Course of Real World Physical Activity and Upper Limb Use After Stroke
Brief Title: Predicting Real World Physical Activity and Upper Limb Use After Stroke
Acronym: REUSE
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01070
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: Physical Activity; Upper Extremity; Movement Sensors; Prognosis; Observational Cohort Study
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment of real world performance
  Interventions: Behavioral: Real world performance of physical activity and arm use

INTERVENTIONS:
Behavioral: Real world performance of physical activity and arm use — Patients will be assessed by using movement sensors and standard clinical assessments

SUMMARY:
Poststroke recovery mainly takes place within the first weeks to months and about 95% of the patients reach their maximum recovery 3 months after stroke onset. Poststroke rehabilitation is initiated as early as possible and aims to reduce functional consequences of stroke, allowing patients to integrate into the community. However, up to 75% of the patients remain disabled in the long term. Strikingly, about 20 to 30% of the patients show functional decline (i.e., learned-nonuse) in the long term - most often after having finished their intensive rehabilitation period - and even stroke survivors who have little or no residual disability are less physically active when compared to their age-matched peers.

Poststroke outcomes can be well predicted early after stroke. However, the deficits early after stroke and the outcomes are measured by standardized clinical tests performed in the laboratory. The drawback of these tests is that they provide information about the best possible abilities of the patients, as they are encouraged by therapists in testing situations. This so called "capacity" does not necessarily reflect what patients do in daily life situations (i.e., "performance" or "real world use").

With the growing interest in the patients' performance, various assessments that objectively measure activities in daily life situations have been developed in the last few years. These devices capture movement in daily life situations in a sensitive and objective way. An additional benefit is that they are less hampered by floor or ceiling effects when compared to clinical laboratory measurements (i.e., clinimetrics). Nevertheless, outcome of real world performance is hardly ever used in clinical trials aiming to determine the effectiveness of stroke rehabilitation interventions. Actually, until today, the natural course of performance remains largely unknown, as are predictors for this course. It is also unknown to which extend patients' subjective reporting of performance matches objectively measured performance. Finally, although it is believed that there is a threshold for, for example, real life use of the paretic arm and further improvement, there is no evidence as to what this threshold is in terms of clinical laboratory measurements.

The present prospective longitudinal cohort study fills in the gap regarding knowledge about the profile and predictability of two performance outcomes during the first year poststroke: engagement in physical activities and the use of the paretic upper limb. In addition, it will provide insight in how physical activity engagement and upper limb use measured by daily life assessments relate to standard clinical laboratory assessments. This knowledge is a prerequisite for the identification of patients' phenotypes and a first essential step towards the development of tailored (i.e., precision medicine), innovative rehabilitation interventions which enhance performance in terms of physical activities or upper limb use in daily life. The ultimate goal is to reduce poststroke disability and associated costs.

RE-USE is a prospective longitudinal observational cohort study of 120 first-ever stroke patients, who will be assessed 3, 10, 28, 90 and 365 days after stroke onset, as well as at discharge of the rehabilitation center.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic or hemorrhagic stroke, confirmed by MRI-DWI and/or CT (recurrent strokes are allowed when already included in this study after a first-ever stroke)
* Paresis or paralysis of the arm and/ or leg
* Living independently before stroke (mRS >2)
* Age 18 years or older
* Written informed consent of the patient or its legal representative after participants' information

Exclusion Criteria:

* Contra-indications on ethical grounds (vulnerable persons)
* Neurological or other diseases affecting upper limb use and/ or physical activity before stroke
* Known or suspected non-compliance, drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Daily life assessment of physical activity engagement and upper limb use | 90 days after stroke onset
  Real world performance, measured with movement sensors (number)

SECONDARY OUTCOMES:
Neurological impairments | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  National Institutes of Health Stroke Scale (0-42 points, lower scores being better)
Upper limb motor function | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Fugl-Meyer Assessment (0-66 points, higher scores being better)
Motor function | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Motricity Index (0-200 points, higher scores being better)
Trunk ability | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Trunk Control Test (0-100 points, higher scores being better)
Sitting and standing balance | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Berg Balance Scale (0-56 points, higher scores being better)
Walking ability (independence) | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Functional Ambulation Categories (0-5 points, higher scores being better)
Gait speed and cadence (time) | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Ten-Meter Walk Test
Upper limb capacity | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Action Research Arm Test (0-56 points, higher scores being better)
Upper limb capacity dexterity | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Box and Block Test (number of blocks)
Global disability | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Modified Rankin Scale (0-6 points, lower scores being better)
Fatigue | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Fatigue Severity Scale (9-63 point, lower scores being better)
Cognition | 3 and 90 days after stroke onset
  Montreal Cognitive Assessment(0-30 points, higher scores being better)
Neglect | 3 and 90 days after stroke onset
  Apples Test (number)
Patient-reported physical activity | 90 and 365 days after stroke onset
  International Physical Activity Questionnaire (3 levels higher levels are better)
Patient-reported daily life upper limb use | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Motor Activity Log - 14 item version (0-5 points, higher scores being better)
Patient-reported changes | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Global Rating of Perceived Changes (1-7 points, higher scores being better; 1-10 points, lower scores being better)
Concomitant movement therapy | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Intensity of therapy based on charts (minutes)
Serious Events and non-serious infections or cardiovascular events | 3, 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Serious Events (1. death; 2. life-threatening illness or injury; 3. in-patient or prolonged hospitalisation; 4. medical or surgical intervention to prevent life threatening illness; 5. led to fetal distress, death or a congenital abnormality or birth defect) and non-serious infections or cardiovascular events
Daily life assessment of physical activity engagement and upper limb use | 3, 10, 28 (expected rehabilitation discharge) and 365 days after stroke onset
  Real world performance, measured with movement sensors (number)
Levels of anxiety and depression | 10, 28, 90 (expected rehabilitation discharge) and 365 days after stroke onset
  Hospital Anxiety and Depression Scale (0-42 points, higher scores indicate greater levels of anxiety or depression)
Health care costs and loss of income | 365 days after stroke onset
  Health care costs and loss of income in relation to the stroke (CHF)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Luft, Prof. Dr., Study Chair — University of Zurich, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey RR, Klaesner JW, Lang CE. Quantifying Real-World Upper-Limb Activity in Nondisabled Adults and Adults With Chronic Stroke. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):969-78. doi: 10.1177/1545968315583720. Epub 2015 Apr 20. PMID 25896988
- [Background] Han CE, Arbib MA, Schweighofer N. Stroke rehabilitation reaches a threshold. PLoS Comput Biol. 2008 Aug 22;4(8):e1000133. doi: 10.1371/journal.pcbi.1000133. PMID 18769588
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Vive-Larsen J, Stoier M, Olsen TS. Outcome and time course of recovery in stroke. Part II: Time course of recovery. The Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 May;76(5):406-12. doi: 10.1016/s0003-9993(95)80568-0. PMID 7741609
- [Background] Kwakkel G, Veerbeek JM, van Wegen EE, Wolf SL. Constraint-induced movement therapy after stroke. Lancet Neurol. 2015 Feb;14(2):224-34. doi: 10.1016/S1474-4422(14)70160-7. PMID 25772900
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Stewart JC, Cramer SC. Patient-reported measures provide unique insights into motor function after stroke. Stroke. 2013 Apr;44(4):1111-6. doi: 10.1161/STROKEAHA.111.674671. Epub 2013 Feb 19. PMID 23422082
- [Background] Stinear CM, Byblow WD. Letter by Stinear and Byblow regarding article, "patient-reported measures provide unique insights into motor function after stroke". Stroke. 2013 Jul;44(7):e79. doi: 10.1161/STROKEAHA.113.001689. Epub 2013 Jun 4. No abstract available. PMID 23735958
- [Background] Taub E, Uswatte G, Mark VW, Morris DM. The learned nonuse phenomenon: implications for rehabilitation. Eura Medicophys. 2006 Sep;42(3):241-56. PMID 17039223
- [Background] Wolfe CD, Crichton SL, Heuschmann PU, McKevitt CJ, Toschke AM, Grieve AP, Rudd AG. Estimates of outcomes up to ten years after stroke: analysis from the prospective South London Stroke Register. PLoS Med. 2011 May;8(5):e1001033. doi: 10.1371/journal.pmed.1001033. Epub 2011 May 17. PMID 21610863
- [Background] Noorkoiv M, Rodgers H, Price CI. Accelerometer measurement of upper extremity movement after stroke: a systematic review of clinical studies. J Neuroeng Rehabil. 2014 Oct 9;11:144. doi: 10.1186/1743-0003-11-144. PMID 25297823
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Derived] Pohl J, Verheyden G, Held JPO, Luft AR, Easthope Awai C, Veerbeek JM. Construct validity and responsiveness of clinical upper limb measures and sensor-based arm use within the first year after stroke: a longitudinal cohort study. J Neuroeng Rehabil. 2025 Jan 29;22(1):14. doi: 10.1186/s12984-024-01512-9. PMID 39881332